CLINICAL TRIAL: NCT00362466
Title: An Open-Label Randomized Phase III Study of Dasatinib vs. High-Dose (600 mg) Imatinib Mesylate in the Treatment of Subjects With Chronic Phase Philadelphia Chromosome-Positive Chronic Myeloid Leukemia Who Are Imatinib Failures or Who Have Had a Suboptimal Response After 3-18 Months of Therapy With 400 mg Imatinib
Brief Title: A Study of Dasatinib vs. High-Dose Imatinib (600 mg) in Patients With Chronic Phase Chronic Myeloid Leukemia (CML) Who Failed to Achieve Complete Cytogenetic Response After 3-18 Months of Imatinib Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient Enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-044
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Leukemia
Keywords: Leukemia (chronic myeloid leukemia - chronic phase)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 50-180 mg once daily (QD)
  Interventions: Drug: Dasatinib
- B (Active Comparator): 200-800 mg QD
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, Once daily, 5-7 years
  Other Names: Sprycel®
  Arms: A
Drug: Imatinib — Tablets, Oral, Once daily, 5-7 years
  Arms: B

SUMMARY:
The purpose of this clinical research study is to compare the rate of complete cytogenetic response of dasatinib to imatinib therapy at 6 months after randomization in chronic phase CML patients. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years diagnosed with Chronic Phase Philadelphia chromosome positive (CP Ph+) CML who have failed to achieve CCyR after 3-18 months of therapy with imatinib 400 mg
* Treatment initiation with imatinib 400 mg within 6 months of initial CML diagnosis
* Able to tolerate chronic administration of imatinib at the highest dose (400-600 mg) the subject has received in the past
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
* Adequate hepatic and renal function

Exclusion Criteria:

* Eligible and willing to undergo immediate autologous/allogeneic stem cell transplant
* Previous diagnosis of accelerated/blast crisis CML
* Subjects with clonal evolution in Ph+ cells observed in ≥2 metaphases
* Previous documentation of T315I mutation
* Uncontrolled or significant cardiovascular disease
* Serious uncontrolled medical disorder/active infection
* History of significant bleeding disorder unrelated to CML
* Intolerance to imatinib ≥400 mg
* Concurrent malignancies other than CML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (42):
- United States (42):
  - Dr. Marshall Schreeder, Huntsville, Alabama
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Alhambra, California
  - Local Institution, Anaheim, California
  - Local Institution, Beverly Hills, California
  - Local Institution, Fullerton, California
  - Local Institution, La Jolla, California
  - Local Institution, La Verne, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Northridge, California
  - Local Institution, Oxnard, California
  - Local Institution, Redondo Beach, California
  - Local Institution, San Francisco, California
  - Local Institution, Santa Maria, California
  - Local Institution, Stanford, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Jacksonville, Florida
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Kansas City, Kansas
  - Local Institution, Hazard, Kentucky
  - Local Institution, Ann Arbor, Michigan
  - Local Institution, Rochester, Minnesota
  - Local Institution, St Louis, Missouri
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Hackensack, New Jersey
  - Local Institution, Buffalo, New York
  - New York Presbyterian Hospital, New York, New York
  - New York Medical College, Valhalla, New York
  - Local Institution, Durham, North Carolina
  - Local Institution, Cleveland, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Baltimore, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 156 subjects were to be enrolled; however, the attempts were unsuccessful and the study was closed after 3 subjects were enrolled. A fourth subject underwent screening, but was not randomized since the subject did not meet the inclusion criteria.
Groups:
- Dasatinib: 100 mg once daily (QD)
- Imatinib: 600 mg QD
Period: Overall Study
Arm/Group | Dasatinib | Imatinib
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib: 100 mg QD
- Total: Total of all reporting groups
Arm/Group | Dasatinib | Imatinib | Total
Number analyzed (Participants) | 2 | 1 | 3
Age Continuous [Number; unit: Participants]
  30- to 39-years-old | 1 | 0 | 1
  40- to 49-years-old | 1 | 0 | 1
  50- to 59-years-old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Complete Cytogenetic Response (CCyR) Rate at Month 6
Description: Cytogenetic Response (CyR) is based on the prevalence of Philadelphia chromosome positive (Ph+) metaphases among cells in metaphase on a bone marrow sample. The criteria for CCyR is 0% Ph+ metaphases among cells in a bone marrow sample.
Time Frame: Month 6
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Major Molecular Response (MMR) Rates
Description: MMR is defined as a 3-log reduction in BCR-ABL gene transcripts from a standardized baseline. Reductions in BCR-ABL transcripts on logarithmic scale are calculated based on the absolute values expressed as percent of ratio of BCR-ABL gene transcripts to the control gene. In this study,ABL was used as the control gene.
Time Frame: Month 3, Month 6, Month 12, Month 24 and Month 36
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: CCyR Rates
Description: CyR is based on the prevalence of Ph+ metaphases among cells in metaphase on a bone marrow sample. The criteria for CCyR is 0% Ph+ metaphases among cells in a bone marrow sample.
Time Frame: Month 3, Month 12, Month 24 and Month 36
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: Participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Estimate Time to MMR and CCyR
Description: Time to MMR is defined as the time from first treatment dose until measurement criteria are first met for MMR. Time to MMR is computed only for subjects who achieved a MMR. Time to CCyR is defined as the time from first treatment dose until measurement criteria are first met for CCyR. Time to CCyR is computed only for subjects who achieved a CCyR.
Time Frame: throughout the study
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: months
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS=time from randomization until progression or death. Participants who died without progression=progression on date of death. Participants who neither progressed nor died were censored on date of last hematologic assessment. Participants who did not receive study treatment and neither progressed nor died were censored on date of randomization.
Time Frame: at 36 months
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to AEs
Description: An AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a patient or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From 2 weeks prior to randomization through Month 36. At least every 4 weeks until all study-related toxicities resolve to baseline, stabilize, or are deemed irreversible.
Population: All treated participants
Measure: Number; unit: events
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 2 | 1
events
  AEs | 3 | 1
  SAEs | 0 | 0
  AEs leading to Discontinuation | 0 | 0
  Deaths | 0 | 0

7. Secondary Outcome: Duration of CCyR and MMR
Description: Duration of CCyR computed for subjects with CCyR as best response; measured from time the criteria are first met for CCyR until date of progression or death. Duration of MMR computed for subjects with MMR as best response; measured from time the criteria are first met for MMR until date the MMR was first lost, disease progression or death.
Time Frame: Throughout the study
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: months
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Best MMR Rates
Description: MMR is defined as a 3-log reduction in BCR-ABL gene transcripts from a standardized baseline. Reductions in BCR-ABL transcripts on logarithmic scale are calculated based on the absolute values expressed as % of ratio of BCR-ABL gene transcripts to the control gene. In this study, ABL was used as the control gene.
Time Frame: throughout study
Population: This analysis was not done. This study was terminated due to insufficient enrollment.
Measure: Number; unit: participants
Arm/Group | Dasatinib | Imatinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dasatinib | Imatinib
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=2) | Imatinib (N=1)
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypokalemia (Investigations) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to insufficient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.